CLINICAL TRIAL: NCT04755114
Title: İnönü University Faculty of Nursing Lecturer
Brief Title: The Effect of Turkish Music and Comedy Film on Pain, Vital Signs and Cortisol Level in Orthopedic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hatice OLTULUOĞLU, Director, Inonu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: İnonuU
Record Dates: First submitted 2021-02-04; First posted 2021-02-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Physiological Parameter; Acute Pain
Keywords: Saliva cortisol; Pain; Funny Film; Türkish Müsic; Nursing; Vital signs
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Turkish Music Group (Experimental): After the patient introduction form is filled, pain level, blood pressure, pulse and respiratory rate will be evaluated, saliva sample will be taken to determine the cortisol level and pre-test data will be collected (0 min). Immediately after the pre-test evaluations, the music group will be played to the music desired by the patient for 30 minutes. Immediately after the interventions, pain level, vital signs will be evaluated and saliva sample will be taken as a final test (30 minutes). The same procedures will be repeated in the 60th minute after the intervention to determine the duration of the interventions applied.
  Interventions: Other: Turkish Music
- Comedy Film Group (Experimental): fter the patient introduction form is filled, pain level, blood pressure, pulse and respiratory rate will be evaluated, saliva sample will be taken to determine the cortisol level and pre-test data will be collected (0 min). Immediately after the pre-test evaluations,the Comedy film group will watch a comedy movie video. Immediately after the interventions, pain level, vital signs will be evaluated and saliva sample will be taken as a final test (30 minutes). The same procedures will be repeated in the 60th minute after the intervention to determine the duration of the interventions applied.
  Interventions: Other: comedy movie
- Control group (No Intervention): After the patient introduction form is filled, pain level, blood pressure, pulse and respiratory rate will be evaluated, saliva sample will be taken to determine the cortisol level and pre-test data will be collected (0 min).
  Pain level and vital signs will be evaluated and saliva sample will be taken for the final test (30th minute) and follow-up (60th minute) simultaneously with the administration group without any intervention.

INTERVENTIONS:
Other: Turkish Music — Turkish Music;In choosing the music, patients will be asked about their favorite vocalist and music pieces before the procedure. The researcher will then download these music pieces from YouTube and create a 30-minute list and listen to patients.
  Arms: Turkish Music Group
Other: comedy movie — Prior to the research, attention will be paid to the selection of comedy films that do not contain violence, swearing and obscene scenes that may adversely affect patients. Prior to the research, attention will be paid to the selection of comedy films that do not contain violence, swearing and obscene scenes that may adversely affect patients. In the selection of comedy films, the opinions of two experts from Mimar Sinan University, Faculty of Fine Arts, Department of Cinema and Television and İnönü University will be preferred, and the films Kemal Sunal and Şener Şen, one of the actors that Turkish people know closely, laugh most and have settled into their culture, will be preferred.
  Arms: Comedy Film Group

SUMMARY:
The aim of this thesis is; It was planned to determine the effect of Turkish music and comedy films on pain, vital signs and cortisol levels of patients who had orthopedic surgery.

The research is a randomized controlled study. 132 patients who meet the research conditions will be included in the study. Patient Information Form, Numerical Pain Rating Scale, Physiological Parameter Form developed by the researcher will be used for data collection.

DETAILED DESCRIPTION:
Turkish Music and Comedy Film Group Data Collection After the patient introduction form is filled, pain level, blood pressure, pulse and respiratory rate will be evaluated, saliva sample will be taken to determine the cortisol level and pre-test data will be collected (0 min). Immediately after the pre-test evaluations, the music group will be played to the music desired by the patient for 30 minutes, and the comedy film group will be shown a comedy movie video. Immediately after the interventions, pain level, vital signs will be evaluated and saliva sample will be taken as a final test (30 minutes). The same procedures will be repeated in the 60th minute after the intervention to determine the duration of the interventions applied.

Control group Data Collection After the patient introduction form is filled, pain level, blood pressure, pulse and respiratory rate will be evaluated, saliva sample will be taken to determine the cortisol level and pre-test data will be collected (0 min).

Pain level and vital signs will be evaluated and saliva sample will be taken for the final test (30th minute) and follow-up (60th minute) simultaneously with the administration group without any intervention.

Collection of Saliva Samples Salivary cortisol is free cortisol not bound to plasma proteins. Considering that the active cortisol is free cortisol, many studies have used the measurement of cortisol in saliva. In addition, salivary cortisol measurement is considered to be a reliable method for measuring stress, since it can be easily obtained, it does not cause stress because it is not invasive, and it shows strong correlation between plasma cortisol levels.

The concentration of cortisol is at its maximum shortly after waking up in the morning, depending on the circadian rhythm. It then declines gradually throughout the day and reaches its lowest level at night. Salivary cortisol also matches the 24-hour rhythm of plasma cortisol.

Saliva samples will be taken at least one hour after the patients wake up so that the circadian changes in cortisol do not affect the results. In order not to change the cortisol levels, the patients will be informed that they should not take orally, chew any substance such as chewing gum, brush teeth, gargle, or smoke one hour after breakfast. It is recommended to rinse the patient's mouth thoroughly with water for 30 seconds before saliva sampling.

To collect saliva sample; Saliva collection tubes were prepared separately for all measurements. Colored labels were affixed on 1.5 ml eppendorf tubes prepared for each measurement of all groups.

Red labels were affixed to the tube of the Turkish music group, green to the tube of the Konedi movie group, and white to the tube of the control group. Numbers given to the participant and the number of measurements (a = 0 minutes, b = 30 minutes, c = 60 minutes) were written on colored labels. In order to facilitate the salivation process, the participants will be given a hookah mouthpiece (sipsi). Saliva collection will be done using passive flow method.

Saliva samples will be stored in the freezer at -20 ° C in the laboratory of the Faculty of Health Sciences, while preserving the cold chain.

ELIGIBILITY:
Inclusion Criteria:

* Does not have any communication problem that will prevent him from understanding the information given, listening to music, watching movies and expressing the pain level correctly,
* Expressing that he experienced "moderate" or "severe" (4 and above according to the Numerical Rating Scale-SDS) pain after the operation,
* Having been operated under general anesthesia and 24 hours after surgery,
* No complications (severe bleeding, nausea, vomiting, etc.) developed in the early postoperative period,
* Without a chronic cardiovascular and respiratory system disease and hormonal problems
* Patients not receiving steroid therapy will be included in the study.

Exclusion Criteria:

* Those with pain score below 4
* Those who have recently used analgesic medication
* Those who have recently consumed any food or drink

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | 5 months
  Each participant has 60 minutes between pretest and posttest. The first follow-up will be done at the first meeting, the second follow-up in the 30th minute, and the last follow-up at the 60th minute.
  There are 11 points on this scale with numbers between 0-10. The "0" point on the left indicates "no pain", "the point" 10 "on the right indicates" the worst pain imaginable ".

CONTACTS AND LOCATIONS:
Overall Officials: Hatice OLTULUOĞLU, Principal Investigator — Inonu University
Locations (1):
- İnonu Ünıversty, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: references — https://pubmed.ncbi.nlm.nih.gov/31785131/